CLINICAL TRIAL: NCT00281229
Title: Innate and Adaptive Immunity in COPD Exacerbations: Surgical Volunteers
Brief Title: T Lymphocyte Cells in Individuals Experiencing an Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L. Curtis, Professor of Internal Medicine, University of Michigan
Other Study IDs: 1328; R01HL082480 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2016-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the lungs of individuals with chronic obstructive pulmonary disease (COPD) contain resident memory T lymphocytes that can produce a combination of cytokines that induce the symptoms of an acute exacerbation of COPD (AE-COPD). Specifically, the study will determine cell-surface receptors of lung T cells in comparison with blood T cells from the same subject, and will examine anti-CD3-activated blood or lung T cells for interleukin (IL)-6 and interferon-gamma production in response to IL-18, and for IL-17A production in response to recombinant IL-23.

DETAILED DESCRIPTION:
BACKGROUND:

COPD is one of the most pressing healthcare problems facing our nation. AE-COPD is responsible for the bulk of healthcare costs, and much of the morbidity and decline in health status among individuals with this common disease. The lack of accepted animal models of AE-COPD necessitates novel approaches using human samples. Advances in the understanding of the pathogenesis have been slowed, in part, due to controversy as to how exacerbations should be defined. The prevailing paradigm has defined AE-COPD as event-based. Such definitions clearly identify groups of patients with accelerated loss of pulmonary function and increased mortality. However, limited data show that symptom-based definitions of AE-COPD also capture episodes inducing significant morbidity and functional decline, and hence of concern to patients. Fundamental mechanisms are lacking to explain AE-COPD defined by either means.

Controversy also surrounds triggers of AE-COPD. Bacteria and viruses are involved in some episodes, but the relative importance of each is intertwined with disputes over the definition of AE-COPD. Progress at linking specific pathogens to molecular pathogenesis has been slow, both due to their diversity, and to the high rates of bacterial colonization of patients with COPD, even in the stable state. Moreover, in many AE-COPD cases, no pathogen can be identified. Without negating the value of analyzing infections with specific species of pathogens, it appears that progress in molecular pathogenesis could be accelerated by focusing on unifying features of the pulmonary immune response during AE-COPD.

DESIGN NARRATIVE:

The research protocol involves isolating lung lymphocytes from surgical specimens of patients already undergoing clinically indicated lung resections. Surgical lung resections may be performed either by open thoracotomy or by video-assisted thoracoscopic surgery (VATS), and could include pneumonectomies, lobectomies, or wedge-excisions, as dictated by clinical care of the patient. This protocol will exclusively use tissue that is of excess after a clinical diagnosis is established. The setting is the operating rooms at the Ann Arbor VA Hospital or the University of Michigan Hospital System. Subjects will be recruited from the outpatient clinics, but will be inpatients at the time of surgery.

Subjects will not undergo any additional procedures beyond routine clinical care as a result of participating in this protocol. However, it is anticipated that the study will have access to the medical record to extract results of demographic data, including occupational exposures and smoking history, pulmonary function testing, and results of imaging and other staging studies.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD AND underwent lung resection for malignancy OR lung volume reduction surgery OR lung transplantation OR lung resection for nodules and masses

Exclusion criteria:

* Mental incompetence or active psychiatric illness
* Currently using more than 20 mg/day of Prednisone
* Asthma as primary clinical pulmonary diagnosis
* Cystic fibrosis
* Clinically significant bronchiectasis
* Other inflammatory or fibrotic lung disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing clinically indicated lung resections.
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2005-09; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
phenotype and in vitro functions of lung lymphocytes | within 3 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Curtis, M.D, Principal Investigator — University of Michigan at Ann Arbor
Locations (2):
- United States (2):
  - University of Michigan at Ann Arbor, Ann Arbor, Michigan
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan

REFERENCES:
- [Background] Freeman CM, Curtis JL, Chensue SW. CC chemokine receptor 5 and CXC chemokine receptor 6 expression by lung CD8+ cells correlates with chronic obstructive pulmonary disease severity. Am J Pathol. 2007 Sep;171(3):767-76. doi: 10.2353/ajpath.2007.061177. Epub 2007 Jul 19. PMID 17640964
- [Background] Curtis JL, Freeman CM, Hogg JC. The immunopathogenesis of chronic obstructive pulmonary disease: insights from recent research. Proc Am Thorac Soc. 2007 Oct 1;4(7):512-21. doi: 10.1513/pats.200701-002FM. PMID 17878463
- [Background] Curtis JL. Cell-mediated adaptive immune defense of the lungs. Proc Am Thorac Soc. 2005;2(5):412-6. doi: 10.1513/pats.200507-070JS. PMID 16322591
- [Result] Freeman CM, Stolberg VR, Crudgington S, Martinez FJ, Han MK, Chensue SW, Arenberg DA, Meldrum CA, McCloskey L, Curtis JL. Human CD56+ cytotoxic lung lymphocytes kill autologous lung cells in chronic obstructive pulmonary disease. PLoS One. 2014 Jul 31;9(7):e103840. doi: 10.1371/journal.pone.0103840. eCollection 2014. PMID 25078269
- [Result] Freeman CM, McCubbrey AL, Crudgington S, Nelson J, Martinez FJ, Han MK, Washko GR Jr, Chensue SW, Arenberg DA, Meldrum CA, McCloskey L, Curtis JL. Basal gene expression by lung CD4+ T cells in chronic obstructive pulmonary disease identifies independent molecular correlates of airflow obstruction and emphysema extent. PLoS One. 2014 May 7;9(5):e96421. doi: 10.1371/journal.pone.0096421. eCollection 2014. PMID 24805101
- [Result] Freeman CM, Martinez FJ, Han MK, Washko GR Jr, McCubbrey AL, Chensue SW, Arenberg DA, Meldrum CA, McCloskey L, Curtis JL. Lung CD8+ T cells in COPD have increased expression of bacterial TLRs. Respir Res. 2013 Feb 1;14(1):13. doi: 10.1186/1465-9921-14-13. PMID 23374856
- [Result] Freeman CM, Han MK, Martinez FJ, Murray S, Liu LX, Chensue SW, Polak TJ, Sonstein J, Todt JC, Ames TM, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Cytotoxic potential of lung CD8(+) T cells increases with chronic obstructive pulmonary disease severity and with in vitro stimulation by IL-18 or IL-15. J Immunol. 2010 Jun 1;184(11):6504-13. doi: 10.4049/jimmunol.1000006. Epub 2010 Apr 28. PMID 20427767
- [Result] Freeman CM, Martinez FJ, Han MK, Ames TM, Chensue SW, Todt JC, Arenberg DA, Meldrum CA, Getty C, McCloskey L, Curtis JL. Lung dendritic cell expression of maturation molecules increases with worsening chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1179-88. doi: 10.1164/rccm.200904-0552OC. Epub 2009 Sep 3. PMID 19729666
- [Result] Freeman CM, Martinez CH, Todt JC, Martinez FJ, Han MK, Thompson DL, McCloskey L, Curtis JL. Acute exacerbations of chronic obstructive pulmonary disease are associated with decreased CD4+ & CD8+ T cells and increased growth & differentiation factor-15 (GDF-15) in peripheral blood. Respir Res. 2015 Aug 5;16(1):94. doi: 10.1186/s12931-015-0251-1. PMID 26243260
- [Derived] Todt JC, Freeman CM, Brown JP, Sonstein J, Ames TM, McCubbrey AL, Martinez FJ, Chensue SW, Beck JM, Curtis JL. Smoking decreases the response of human lung macrophages to double-stranded RNA by reducing TLR3 expression. Respir Res. 2013 Mar 9;14(1):33. doi: 10.1186/1465-9921-14-33. PMID 23497334
- See also: COPD Foundation — http://www.copdfoundation.org/